CLINICAL TRIAL: NCT02579720
Title: Non-interventional Study A Multicentre Observational Study for Revaccination With Pollinex® Quattro in Patients With a Recurrent Grass Pollen Allergy
Brief Title: Revaccination With Pollinex® Quattro
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Ralph Mösges (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Ralph Mösges, Professor, University Hospital of Cologne
Organization: University Hospital of Cologne (Other)
Other Study IDs: BC Grass Booster 01 2014
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Allergic Rhinitis
Keywords: Recurrent Grass Pollen Allergy; Pollinex® Quattro
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Pollinex® Quattro Patients: Patients treated with Pollinex® Quattro
- Group 2: Control Patients: Patients who decided to use only anti-allergic drugs during the grass pollen season

SUMMARY:
The purpose of this non interventional study (NIS) was to observe the efficacy of Pollinex® Quattro as a short-term revaccination in patients who have already been successfully desensitized at least five years ago against grass-pollen but developed a recurrent allergy.

DETAILED DESCRIPTION:
The increasing prevalence of allergies represents a major problem for the health care system. Approximately 500 million people are suffering worldwide from allergic rhinitis (AR). Allergic rhinitis is a Type 1 hypersensitive disorder, initiated by IgE antibodies. Whereas seasonal allergic rhinitis (SAR) is caused by different allergens found outdoors such as grass, tree and weed pollen, perennial allergic rhinitis (PAR) is caused by allergens that are mainly found indoors such as dust mites, mould or animal hair.

Specific immunotherapy (SIT) presently constitutes the only causal therapy available and is common practice. SIT is indicated in cases of IgE-mediated allergic diseases and includes two forms of treatment options: subcutaneous (SCIT) and sublingual immunotherapy (SLIT). Both therapies aim to train the immune system not react to supposed pathological allergens, but instead to develop tolerance to them.

Even though allergy vaccinations have been applied for a century, the commonly used SCIT requires up to 90 injections over three to five years. Pollinex® Quattro is currently the only ultra-short term medicinal product which requires only four preseasonal injections. The immunological effect associated with Pollinex® Quattro shows an increase of allergen-specific IgG antibodies and a decrease of allergen-specific IgE antibodies as well as a shift from a Th2 to a more Th1 type-immune reaction. Previous studies on the therapeutic efficacy of Pollinex® Quattro have come to a positive conclusion in regards to tolerability and decrease of allergic symptoms. As an ultra-short course SCIT, Pollinex® Quattro might decrease the number of noncompliance and withdrawal for revaccination in patients that have already undergone an intensive immunisation therapy.

In this non-interventional study, patients who were treated with Pollinex® Quattro and patients who decided to use anti-allergic drugs for the treatment of their grass pollen allergy were compared due to their allergic symptoms in the grass pollen season from May to July. For this purpose, the rhinoconjunctivitis and asthmatic symptoms as well as the use of concomitant medication were documented in a dia

ELIGIBILITY:
Inclusion Criteria:

* Adults and children from the age of 12 years on, who are diagnosed with recurrent seasonal allergic rhinitis (SAR) caused by grass pollen.

A previous specific immunotherapy finished at least five years ago had to be successful.

Exclusion Criteria:

* Contraindications according to the patient information leaflet

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children from the age of 12 years on, who are diagnosed with recurrent seasonal allergic rhinitis (SAR) caused by grass pollen.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the efficacy of Pollinex® Quattro based on the Combined Symptom and Medication Score (CSMS) (Pfaar et al., 2014). | 3 months
  The CSMS consists of the six individual rhinoconjunctivitis scores for sneezing, rhinorrhoea, nasal pruritus, nasal congestion, ocular pruritus and watery eyes, the asthma scores for cough, breathlessness, wheeze and tightness in the chest as well as the score for the use of concomitant medication (oral antihistamines, nasal corticosteroids, oral corticosteroids, asthma inhalation spray). The symptoms and the use of drugs were documented in a diary: The symptom score was:
  0=none, 1=mild, 2=moderate, 3=severe. Evaluation will be done for the peak of the grass pollen season, defined by those 30 consecutive days per center with the highest local grass pollen counts (according to Deutscher Wetterdienst Medizin-Meteorologie, http://www.dwd.de) measured in the nearest pollen count station in that region.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kramer, Prof. Dr., Study Director — Bencard Allergie GmbH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosewich M, Lee D, Zielen S. Pollinex Quattro: an innovative four injections immunotherapy in allergic rhinitis. Hum Vaccin Immunother. 2013 Jul;9(7):1523-31. doi: 10.4161/hv.24631. Epub 2013 Apr 12. PMID 23584250
- [Result] Pfaar O, Demoly P, Gerth van Wijk R, Bonini S, Bousquet J, Canonica GW, Durham SR, Jacobsen L, Malling HJ, Mosges R, Papadopoulos NG, Rak S, Rodriguez del Rio P, Valovirta E, Wahn U, Calderon MA; European Academy of Allergy and Clinical Immunology. Recommendations for the standardization of clinical outcomes used in allergen immunotherapy trials for allergic rhinoconjunctivitis: an EAACI Position Paper. Allergy. 2014 Jul;69(7):854-67. doi: 10.1111/all.12383. Epub 2014 Apr 25. PMID 24761804